CLINICAL TRIAL: NCT02192905
Title: Feasibility Trial of a Problem-Solving Weight Loss Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Worcester Polytechnic Institute (Other)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-237; 1R21DK098556-01 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-07-17 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral Weight Loss + Habit (Experimental): Participants will receive 8 week of an online-delivered weight loss intervention adapted from the Diabetes Prevention Program Lifestyle Intervention and will use the Habit mobile app during the study.
  Interventions: Behavioral: Diabetes Prevention Program Lifestyle Intervention

INTERVENTIONS:
Behavioral: Diabetes Prevention Program Lifestyle Intervention

SUMMARY:
The purpose of this research was to develop and test the feasibility of Habit, a weight loss mobile application that was designed to coach patients through their weight loss challenges. In a pilot trial in 43 obese participants, investigators tested the feasibility of the Smart Coach mobile application when paired with a shortened online-delivered (8-week) behavioral weight loss intervention. Feasibility outcomes included frequency and duration of usage of the mobile app and each feature, recruitment, and retention. Post-intervention focus groups discussed the feasibility and acceptability of the intervention. The investigators also performed exploratory analyses comparing conditions on problem solving skills and weight loss at 8 and 16 weeks, which will inform a subsequent randomized controlled efficacy trial.

DETAILED DESCRIPTION:
The investigators developed and tested the feasibility of Habit, a weight loss mobile app that includes common features such as self-monitoring, goal setting, and a social network, but even more importantly, an avatar-facilitated, idiographic problem solving feature that processes information intelligently to help patients identify solutions to their weight loss problems. In a pilot trial in 43 obese participants, investigators tested the feasibility of the Habit mobile application when paired with a shortened (8 week) behavioral weight loss intervention. Feasibility outcomes included frequency and duration of usage of the mobile app and each feature, recruitment, and retention. The investigators also performed analyses on problem solving skills and weight loss at 8 and 16 weeks, which will inform a subsequent randomized controlled efficacy trial. Data will support an efficacy trial of a Habit-assisted brief behavioral weight loss intervention relative to a brief behavioral weight loss intervention alone with 1 year follow-up. The investigators overarching goal is to develop mobile technology that reduces the intensity of lifestyle interventions as far as possible while preserving weight loss outcomes, to ultimately broaden reach.

ELIGIBILITY:
Inclusion: Participants must 1) have a BMI between 30 and 45, 2) currently uses a smartphone with Android software, 3) have connectivity to the internet at home and work, 4) have PCP written clearance, and 5) age 18 or older.

Exclusion:

1. Ages <18
2. BMI <30 and >45
3. Does not currently use a smart phone with Android software version 4.4 or later
4. Does not use a smartphone supported by the app (will assess model and type of phone for each participant)
5. Does not have connectivity to the internet at home and work; or wifi access at home
6. Does not use smart phone regularly throughout the day
7. Has not used Android smartphone for at least a year
8. Has not used a weight loss mobile app in the last 6 months
9. Does not have a Facebook account, uses it infrequently, or does not actively engage on Facebook
10. Does not have a gmail account or is unwilling to create one
11. Does not have PCP written clearance
12. Bipolar disorder, substance abuse, psychosis, bulimia, or severe depression
13. Pregnant or lactating
14. Had bariatric surgery
15. Medication affecting weight
16. Adults unwilling to provide consent
17. Prisoners
18. Unable to read or understand English
19. Has type 1 or 2 diabetes
20. Have concerns about being audiotaped
21. Unable to walk unaided
22. Has any medical condition that precludes lifestyle changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Pagoto S, Tulu B, Agu E, Waring ME, Oleski JL, Jake-Schoffman DE. Using the Habit App for Weight Loss Problem Solving: Development and Feasibility Study. JMIR Mhealth Uhealth. 2018 Jun 20;6(6):e145. doi: 10.2196/mhealth.9801. PMID 29925496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to begin the intervention, participants needed to complete: an online eligibility screener, a telephone screening, the consent process, a screening survey, medical clearance, and a webinar. Missing any of these components would be reason for exclusion.
Groups:
- Behavioral Weight Loss + Habit: Individuals randomized to this condition will receive 8 weeks of an online-delivered weight loss intervention adapted from the Diabetes Prevention Program Lifestyle Intervention and will use the Habit mobile app during the study.
  Diabetes Prevention Program Lifestyle Intervention
Period: Overall Study
Arm/Group | Behavioral Weight Loss + Habit
Started | 43
Completed | 42 (Reporting a minimum of current weight at 16-week follow-up)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.33 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 35
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43
Weight [Mean (Standard Deviation); unit: pounds] | 202.02 (42.6)
Social-Problem Solving Inventory-Revised [Mean (Standard Deviation); unit: Total score] — The social problem solving inventory measures strengths and weaknesses in ability to solve problems. The measure includes sub scales (positive problem orientation, rational problem-solving, negative problem orientation, impulsivity/carelessness style, and avoidance style). The means of the subscales are summed and then matched against an age chart to achieve the total score for the age being studied. This is done for each participant. The total score is being reported in these results. The scoring range includes 28 to 140. The higher the score the higher the problem solving ability.
  Total score | 107.3 (14.75)
Facebook Use [Count of Participants; unit: Participants]
  Uses Facebook 5-6 times per week | 9
  Uses Facebook daily or more | 34

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Total Uses)
Description: Mean total uses of the problem solving function of the mobile application
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: mean uses of the app
Groups:
- Behavioral Weight Loss + Habit: Participants will receive 8 weeks of an online-delivered weight loss intervention adapted from the Diabetes Prevention Program Lifestyle Intervention and will use the Habit mobile app during the study.
  Diabetes Prevention Program Lifestyle Intervention
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
mean uses of the app | 23.7 (19)

2. Primary Outcome: Feasibility (Total Habits Attempted)
Description: Total amount of new habits attempted during the study
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: mean habits attempted
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
mean habits attempted | 17.4 (11.6)

3. Primary Outcome: Feasibility (Recruitment Rates)
Description: Recruitment rates include the total number of participants contacting us to participate, which includes the intervention participants plus those screened out prior to starting the intervention (Total screened = 559; Total intervention participants = 43)
Time Frame: Baseline
Population: Of the total number of participants screened for this study (n=559), 7.69% (n=43) were enrolled into the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 559
Participants | 43

4. Primary Outcome: Feasibility (Retention Rates)
Description: Total attendance at groups and total withdrawn from the study
Time Frame: 8-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
Participants | 42

5. Secondary Outcome: Problem Solving Inventory
Description: The social problem solving inventory measures strengths and weaknesses in ability to solve problems in all areas of life. The measure includes sub scales (positive problem orientation, rational problem-solving, negative problem orientation, impulsivity/carelessness style, and avoidance style). The means of the subscales are summed and then matched against an age chart to achieve the total score for the age being studied. This is done for each participant. The scoring range is 28 to 140. The higher the score the higher the problem solving ability.The change from baseline to 8-weeks is calculated by subtracting the baseline score from the 8 week score and then doing a 1-sample t-test of whether or not the change was different than 0.
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
Total score | -.64 (8.31)
Statistical Analysis 1: Comparison: Behavioral Weight Loss + Habit; Test type: Other — One-sample t-test testing the mean positive problem solving change from baseline to week 8; p = .63, t-test, 2 sided; Mean Difference (Final Values) = -.64, 95% CI 2-sided [-3.34 to 2.05], Standard Deviation 8.31

6. Secondary Outcome: % Weight Change
Description: Measured in pounds with a digital scale
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: percentage of pounds
Groups:
- Behavioral Weight Loss + Habit: Individuals randomized to this condition will receive 8 week of an online-delivered weight loss intervention adapted from the Diabetes Prevention Program Lifestyle Intervention and will use the Habit mobile app during the study.
  Diabetes Prevention Program Lifestyle Intervention
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
percentage of pounds | -1.9 (3.0)
Statistical Analysis 1: Comparison: Behavioral Weight Loss + Habit; Test type: Other — One-sample t-test testing the mean within-person percent weight change from baseline to week 8; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -.019, 95% CI 2-sided [-.0285 to -.0096], Standard Deviation .03

7. Secondary Outcome: % Weight Change
Description: Measured in pounds with a digital scale
Time Frame: 16 week follow-up
Measure: Mean (Standard Deviation); unit: percentage of pounds
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
percentage of pounds | -1.67 (7.3)
Statistical Analysis 1: Comparison: Behavioral Weight Loss + Habit; Test type: Other — One-sample t-test testing the mean within-person percent weight change from baseline to week 16; p = 0.143, t-test, 2 sided; Mean Difference (Final Values) = -.017, 95% CI 2-sided [-.039 to .006], Standard Deviation .011

8. Secondary Outcome: Social Problem Solving Inventory
Description: The social problem solving inventory measures strengths and weaknesses in ability to solve problems in all areas of life. The measure includes sub scales (positive problem orientation, rational problem-solving, negative problem orientation, impulsivity/carelessness style, and avoidance style). The means of the subscales are summed and then matched against an age chart to achieve the total score for the age being studied. This is done for each participant. The scoring range is 28 to 140. The higher the score the higher the problem solving ability. The change from baseline to 16-weeks is calculated by subtracting the baseline score from the 16 week score and then doing a 1-sample t-test of whether or not the change was different than 0.
Time Frame: 16-week follow-up
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Behavioral Weight Loss + Habit
Number analyzed (Participants) | 43
Total score | -.76 (13.07)
Statistical Analysis 1: Comparison: Behavioral Weight Loss + Habit; Test type: Other — One-sample t-test testing the mean positive problem solving change from baseline to week 16; p = .73, t-test, 2 sided; Mean Difference (Final Values) = -.76, 95% CI 2-sided [-5.11 to 3.6], Standard Deviation 13.07

ADVERSE EVENTS:
Time Frame: Participants were in the study for 16 weeks and were monitored for the occurrence of adverse events throughout the study. Adverse events were documented during the interventions, at the 8-week assessment, and the 16-week assessment.
Arm/Group | Behavioral Weight Loss + Habit
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 9/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Weight Loss + Habit (N=43)
Cold, flu, or virus (General disorders) | 6 (6)
Previous condition worsening (General disorders) | 2 (2)
Injury (General disorders) | 1 (1) — Injured back while cleaning

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No